CLINICAL TRIAL: NCT01585233
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Sequential, Multiple Dose Escalation Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of ASKP1240 in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Multiple Dose Escalation Study of ASKP1240 in Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7163-CL-0107
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis
Keywords: Moderate Psoriasis; Severe Psoriasis; Skin disease; ASKP1240; CD40 antigen; Anti-CD40 monoclonal antibody
MeSH Terms: conditions — Psoriasis; Skin Diseases | interventions — bleselumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): ASKP1240 lowest dose
  Interventions: Drug: ASKP1240
- Cohort 2 (Experimental): ASKP1240 low dose
  Interventions: Drug: ASKP1240
- Cohort 3 (Experimental): ASKP1240 high dose
  Interventions: Drug: ASKP1240
- Cohort 4 (Experimental): ASKP1240 highest dose
  Interventions: Drug: ASKP1240
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASKP1240 — Intravenous
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: Placebo — Intravenous
  Arms: Placebo

SUMMARY:
The purpose of this study is to explore the safety and tolerability of multiple doses of ASKP1240 compared to placebo and determine Pharmacokinetics and Pharmacodynamics in subjects with moderate to severe psoriasis.

DETAILED DESCRIPTION:
Treatment with ASKP1240 or placebo will be over 4 weeks (Baseline/Day 1, Days 15 and Day 29) with 12 weeks of follow-up for a total of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a clinical diagnosis of moderate to severe plaque psoriasis for 6 months or longer with at least 5% or greater Body Surface Area (BSA) affected with plaque psoriasis
* Subject must be a candidate for phototherapy and/or systemic therapy
* Subject must agree to avoid prolonged exposure to the sun and avoid the use of tanning booths or other ultraviolet light sources during the study
* Female subject must be either:

  * post-menopausal (defined as at least 1 year without any menses) prior to Screening, or
  * premenarchal prior to Screening, or
  * documented surgically sterile or status post hysterectomy (at least 1 month prior to Screening), or
* if of childbearing potential, must have a negative serum pregnancy test at Screening and if sexually active must be using highly effective contraception. All sexually active subjects will be required to use highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at Screening and throughout the study period and for 28 days [or 5 five half lives of the study drug whichever is longer] after final study drug administration.
* Female subject must not be lactating and must not be breastfeeding at Screening or during the study period and for 28 days [or 5 five half lives of the study drug whichever is longer] after final study drug administration.
* Female subject must not donate ova starting at Screening and throughout the study period and for 28 days [or 5 five half lives of the study drug whichever is longer] after final study drug administration.
* Male subject and their female spouse/partners who are sexually active must be using highly effective contraception1 consisting of two forms of birth control (one of which must be a barrier method) starting at Screening and continue throughout the study period and for 28 days [or 5 five half lives of the study drug whichever is longer] after final study drug administration.
* Male subject must not donate sperm starting at Screening and throughout the study period and for at least 28 days [or 5 five half lives of the study drug whichever is longer] after final study drug administration.
* Highly effective contraception is defined as:

  * Established use of oral, injected or implanted hormonal methods of contraception.
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * Barrier methods of contraception: Condom alone or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
* Subject must be willing and able to comply with the study requirements, including prohibited concomitant medication restrictions.
* Waivers to the inclusion criteria will NOT be allowed.

Exclusion Criteria:

* Subject has non-plaque psoriasis (such as guttate, erythrodermic or pustular psoriasis)
* Subject has received treatment with systemic, non-biologic psoriasis therapy or other systemic immunosuppressant including investigational use of an approved agent within the last 30 days or 5 half-lives, whichever is longer, prior to the first dose of study drug
* Subject has ever been treated with efalizumab (Raptiva®)
* Subject has a total B lymphocyte count by flow cytometric determination that is less than the lower limit of normal
* Subject has a hemoglobin, that are below the lower limit
* Subject has a total white count, total lymphocyte count, total neutrophil count or total platelet that are below the lower limit
* Subject has any of the following lab values:

  * ALT ≥ 1.5 x upper limit of normal
  * AST ≥ 1.5 x upper limit of normal
  * Total bilirubin ≥ 1.5 x upper limit of normal
* Subject has previously received ASKP1240 or has participated in a study involving ASKP1240
* Subject has > 45 body mass index (BMI)
* Subject with a positive Tubercle Bacillus (TB) test who has not previously received adequate antimicrobial therapy for TB or is currently on, or is planned to start TB antimicrobial therapy
* Subject has abnormal chest x-ray indicative of acute or chronic lung disease
* Subject has uncontrolled intercurrent illness, including, but not limited to ongoing or active infection, any clinically significant cardiac disease seizure disorder, or psychiatric illness/social situations that would limit compliance with study requirements
* Subject has a history of any malignancy regardless of the location and the time of diagnosis in the last 5 years (including in-situ carcinoma of the cervix, but excluding successfully treated non-metastatic basal cell and squamous cell carcinoma)
* Subject has received live or live attenuated virus vaccinations within the last 30 days prior to first dose of study drug
* Subject has received treatment with another investigational drug within 30 days or 5 half-lives; whichever is longer, prior to the initiation of Screening
* Subject has a positive test for hepatitis B surface antigen (HBsAg) or hepatitis C (HCV) antibody
* Subject has a history of a positive test for human immunodeficiency virus (HIV) infection
* Subject has received treatment with systemic, biologic psoriasis therapy or other systemic immunosuppressant including investigational use of an approved agent within the last 56 days or 5 half-lives whichever is longer, prior to the first dose of study drug
* Waivers to the exclusion criteria will NOT be allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2015-01-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of ASKP1240: Area under the curve 0-336 (AUC336 ) | Day 1 to Day 113 (12 visits)
Pharmacokinetics of ASKP1240: Maximum Concentration (Cmax) | Day 1 to Day 113 (12 visits)
Pharmacodynamic variable: CD40 receptor occupancy on peripheral blood B cells | Day 1 to Day 113 (12 visits)
Characterize safety profile of ASKP1240 through adverse event reporting, vital signs, clinical laboratory evaluations, physical examinations and 12-lead electrocardiograms (ECGs) | 113 Days

SECONDARY OUTCOMES:
Mean change from baseline to 8 weeks in Psoriasis Area Severity Index (PASI) score | Baseline and 8 weeks
Mean change from baseline to 8 weeks in Physicians Static Global Assessment (PSGA) score | Baseline and 8 weeks
Proportion of Subjects Achieving Treatment Success | 8 weeks
  Success of the treatment of psoriasis is defined as a score of 1 (almost clear) or 0 (clear) as measured by the PSGA
Mean change from baseline to 8 weeks in % Body Surface Area (BSA) | Baseline and 8 weeks
Cytokine Concentration | Day 1 to Day 113 (9 visits)
Anti-ASKP1240 antibodies | Day 1 to Day 113 (8 visits )
Lymphocyte subset quantitation | Day 1 to Day 113 (9 visits)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development
Locations (13):
- Australia (4):
  - Specialist Connect, Brisbane, Queensland
  - CMAX, Adelaide, Victoria
  - Epworth Hospital, Richmond, Victoria
  - Linear Research, Nedlands, Western Australia
- Canada (5):
  - Durondel C.P. Inc, The Dermatology Clinic, Moncton, New Brunswick
  - New Lab Clinical Research, St. John's, Newfoundland and Labrador
  - Ultranova Skincare, Barrie, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Innovaderm Research, Inc., Montreal, Quebec
- New Zealand (4):
  - Auckland Clinical Studies, Auckland
  - Christchurch Clincial Studies Trust, Ltd., Christchurch
  - P3 Research, Tauranga, Tauranga
  - P3 Research, Wellington, Wellington

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency.

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=25563&tenant=MT_AST_9011